CLINICAL TRIAL: NCT06108635
Title: Additional Effects of Maitland Mobilization With Mckenzie Exercises on Kinesiophobia and Range of Motion in Upper Cross Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUI/CTR/2023/19
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: Parallel Group Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: A single blinded study will be used in which data analyzer will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): McKenzie exercises with moist heat therapy will be given as intervention to experimental group. 2 sets of 5 reps will be given then progressed to 3 sets of 10 repetitions .Participants will be given Hot pack for 15 minutes.
  Interventions: Procedure: McKenzie Exercises; Procedure: Heat Therapy
- Group B (Experimental): The patients will be given Maitland mobilization (central glide on effected cervical spinous process) with McKenzie exercises. Grade i and ii mobilizations will be given in week 1 and then progressed to grade iii and iv in week 2. The total time duration will be 25-30 minutes. Participants will be given Hot pack for 15 minutes.
  Interventions: Procedure: McKenzie Exercises; Procedure: Maitland mobilization; Procedure: Heat Therapy

INTERVENTIONS:
Procedure: McKenzie Exercises — These can be performed in sitting and the protocol includes,
  1. Retraction and extension
  2. Retraction and extension with rotation
  3. Postural correction
  There will be 2 sets of 5 repetitions in week 1 and 3 sets of 10 repetitions in week 2 followed by alternative days in a week. Each set is 30 seconds and each repetition is given in 2 seconds.
Procedure: Maitland mobilization — The grade I and II Maitland mobilizations are given in week 1 and then progressed to grade III and IV in week 2
  Arms: Group B
Procedure: Heat Therapy — Moist heat therapy with hot pack.

SUMMARY:
Upper cross syndrome is a postural condition that is characterized by muscle imbalance in neck region. It is described as a pattern of crossed tightness in trapezius, levator scapulae and pectoralis major and minor with crossed weakness in neck flexors,rhomboids,serratus anterior weakness due to poor working habits and inappropriate ergonomics. It has multiple treatment options and manual therapy is on of them. Maitland mobilizations are widely used for upper cross syndrome. However limited literature is available on the additional effects of Maitland mobilizations with Mckenzie exercises in upper cross syndrome.

DETAILED DESCRIPTION:
Upper cross syndrome is a postural condition that is experinced by 32.43% in desk workers. It is one of the most prevelant leading cause of neck pain and musculoskeletal conditions that has a major impact on a person life by effecting activities of daily living.Neck pain ranked 21st among Global burden of diseses and fourth highest overall for all disabilities. Prevelance of neck pain in Pakistan is 62%. Neck pain has a strong positive correlation with kinesiophobia. Kinesiophobia is a strong predictor of pain intensity,proprioception and functional performance. Patients with upper cross syndrome presents with forward head posture, protracted and elongated shoulders,khyphosis of thoracic spine,winging of scapula and decreased thoracic spine mobility. Upper cross syndrome occurs due to poor faulty posture, extensive use of mobile,laptops,watching T.V,driving and all the other activities that encourages this postural stance.

This study will be a Randomized Control Trial conducted in rehab opd of Fauji Foundation hospital. Both genders with age 18-45 years who had diagnosed with upper cross syndrome will be recruited into two groups using non probability purposive sampling technique. Sample size has been calculated by using open epi sample calculator and it is calculated to be 28. Patients with primary neck pain complain referred to rehab opd of FFH and local physiotherapy clinics of Rawalpindi/Islamabad will be recruited according to the eligibility criteria. Participants will be briefed regarding study objectives, study procedures, risks and benefits of treatment, voluntarily participation and right to withdraw. After taking informed consent,basic demographics, baseline assessment, participants will be randomly allocated into the two groups using sealed enveloped method. Group A(controlled group) will be recieving moist heat therapy(15 minutes hot pack) and Mckenzie exercise(5 reps x 2 sets in week 1 then progressed to 10 reps x 3 sets in week 2) . While group B will be given Maitland mobilization (Central glidewith grade i and ii mobilizations in week 1 and then progressed to grade iii and iv in week 2) with Mckenzie exercises along with moist heat therapy. Before and after the intoduction of intervention kinesiophobia,range of motion and pain will be assessed before and after the treatment.Frequency: thrice biweekly for 2 weeks for a total of 6 treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age group:18-45 years with diagnosed upper cross syndrome
* Both males and females
* Neck pain with a score between 4-8 in NPRS
* Able to provide informed consent and understand therapists instruction

Exclusion Criteria:

* History of Cervical or upper limb fracture
* Vertibrobasilar insufficiency
* Cervical spine surgery
* Spinal infections and tumors
* Osteoporosis
* Metabolic disorders
* Rheumatiod Arthritis
* Inflammatory Arthritis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 2 weeks
  It will be defined as an excessive irrational and debilitating fear of movement and is associated with a feeling of vulnerability to injury in response to movement and includes more than 20 score on Tampa scale of kinesiophobia.
Range of motion | 2 weeks
  It is composed of three inclinometers in frontal, sagittal and horizontal position. Each compass of the inclinometer is placed on the zero degree and measures the range of motion.

SECONDARY OUTCOMES:
Severity of neck pain | 2 weeks
  Numeric pain rating scale. Greater score means greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan